CLINICAL TRIAL: NCT05632549
Title: The Possible Efficacy and Safety of L-carnitine and Biotin as Adjunctive Therapies in Children With Moderate Persistent Asthma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed osama khedr, Clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35652/8/22
Record Dates: First submitted 2022-11-10; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Moderate Persistent Asthma
MeSH Terms: interventions — Carnitine; Tablets; Biotin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Group 1 (n=22) which will receive traditional therapy plus placebo capsule twice daily for 3 months.
  Interventions: Drug: Placebo
- L-carnitine (Experimental): Group 2 (n=22) which will receive traditional therapy plus L-carnitine capsules (500 mg twice daily) for 3 months.
  Interventions: Drug: L-Carnitine 500Mg Oral Tablet
- Biotin (Experimental): Group 3 (n=22) which will receive traditional therapy plus Biotin capsules (5 mg twice daily) for 3 months.
  Interventions: Drug: Biotin Capsules

INTERVENTIONS:
Drug: Placebo — Group 1 (n=22) which will receive traditional therapy plus placebo capsule twice daily for 3 months.
  Arms: Placebo
Drug: L-Carnitine 500Mg Oral Tablet — Group 2 (n=22) which will receive traditional therapy plus L-carnitine capsules (500 mg twice daily) for 3 months.
  Arms: L-carnitine
Drug: Biotin Capsules — Group 3 (n=22) which will receive traditional therapy plus Biotin capsules (5 mg twice daily) for 3 months.
  Arms: Biotin

SUMMARY:
The Possible Efficacy and Safety of L-carnitine and Biotin as Adjunctive Therapies in Children with Moderate Persistent Asthma

ELIGIBILITY:
Inclusion Criteria:

* Children with moderate persistent asthma
* Age range of 8-< 18 years old
* Both sex

Exclusion Criteria:

* Children with any pulmonary or chronic systemic diseases other than asthma (cystic fibrosis, bronchiectasis, tuberculosis, diabetes mellitus, and liver disease).
* Children with immunodeficiency.
* Children with thyroid disorder.
* Children with recent infection (especially pneumonia), surgery, anesthesia.
* Children having clinical evidence of any heart renal and hepatic diseases.
* Children having cystic fibrosis or congenital respiratory disease.
* Children having chronic diarrhea and mal-absorption.
* Children having clinical evidence of malnutrition.
* Children on medications that could interfere with L-carnitine level including antibiotics use. (particularly ampicillins) and anti- convulsing particularly valoproic acid.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-08-08 (Estimated); Study Completion 2024-08-08 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function test (PFT) | 3 months
  Pulmonary Function Test (PFT) using a calibrated computerized spirometer. Subjects will be submitted to 3 acceptable Forced Vital Capacity (FVC) maneuvers according to American Thoracic Society recommendations (NIH, 2007). The maximum percentage in Forced Expiratory Volume in 1 second (FEV1) value from 3 readings will be calculated.
Childhood asthma control test (C-ACT) | 3 months
  Childhood-Asthma Control Test (C-ACT) is a 7-item child- and caregiver-completed tool with a scoring range of 0-27. The higher scores indicate better control. A score of 19 or less indicates that the asthma is not well controlled.

SECONDARY OUTCOMES:
serum levels of TGF-β1 | at baseline and 3 months after intervention
  the change in serum levels of TGF-β1
serum levels of TNF-α | at baseline and 3 months after intervention
  Change in serum level of TNF-α
serum levels of 8-OHDG | at baseline and 3 months after intervention
  the change in serum levels of 8-OHDG

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt